CLINICAL TRIAL: NCT05281874
Title: Personalized Integrated Alcohol and Sexual Assault Prevention Among College Students
Acronym: +Change
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Amanda Gilmore, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GeorgiaSU
Record Dates: First submitted 2021-11-05; First posted 2022-03-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and principal investigator will be masked to intervention conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): A healthy lifestyles attention control will be used as the control condition. We will match the control and intervention conditions on content (text, pictures, number of pages); type (interactive vs. psychoeducation); and average completion time.
  Interventions: Behavioral: A healthy lifestyles attention control
- Positive Change (+Change) (Experimental): This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse and sexual assault. It targets alcohol, sexual assault victimization risk, sexual assault perpetration, and bystander intervention. It is tailored by gender and sexual orientation.
  Interventions: Behavioral: Positive Change (+Change)
- Positive Change (+Change) Plus Booster (Experimental): This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse and sexual assault. It targets alcohol, sexual assault victimization risk, sexual assault perpetration, and bystander intervention. It is tailored by gender and sexual orientation. It is provided at baseline and a booster at 6 months.
  Interventions: Behavioral: Positive Change (+Change) Plus Booster

INTERVENTIONS:
Behavioral: Positive Change (+Change) — This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse and sexual assault. It targets alcohol, sexual assault victimization risk, sexual assault perpetration, and bystander intervention. It is tailored by gender and sexual orientation.
  Arms: Positive Change (+Change)
Behavioral: A healthy lifestyles attention control — A healthy lifestyles attention control will be used as the control condition. We will match the control and intervention conditions on content (text, pictures, number of pages); type (interactive vs. psychoeducation); and average completion time.
  Arms: Control
Behavioral: Positive Change (+Change) Plus Booster — Positive Change (+Change) Plus Booster
  Arms: Positive Change (+Change) Plus Booster

SUMMARY:
Heavy episodic drinking and sexual assault are problematic on college campuses. This study includes a randomized controlled trial of Positive Change (+Change), an integrated alcohol and sexual assault prevention program, compared to an attention-matched control condition across two universities in reducing alcohol use, sexual assault victimization, sexual assault perpetration, and increasing sexual assault bystander intervention. This study will also test the efficacy of +Change plus Booster session, an identical version of +Change delivered 6 months after the baseline, compared to +Change alone in long-term reductions in alcohol use, sexual assault victimization, sexual assault perpetration, and increases in sexual assault bystander intervention. This research is the next step of a NIAAA-funded planning grant (R34AA025691).

DETAILED DESCRIPTION:
Aim 1: Test the efficacy of Positive Change (+Change) among college students in each risk group (cisgender heterosexual men; cisgender heterosexual women; LGBTQ). Students aged 18-25 who engage in heavy episodic drinking will be recruited from 2 large public universities (n = 3,300) and will be randomly assigned to +Change, +Change plus +Booster, or an attention control. Alcohol use, sexual assault (victimization and perpetration), and bystander intervention will be assessed at baseline, 3-, 6-, 9-, and 12-month follow-ups.

H1a: +Change conditions (+Change and +Change plus Booster) will result in less alcohol use, less sexual assault (victimization and perpetration), and more bystander intervention compared to the control condition at 3-month follow-up and maintained at 6 months.

H1b: +Change plus booster at 6-months will maintain less alcohol use, less sexual assault (victimization and perpetration), and more bystander intervention compared to +Change over 9- and 12-month follow-ups (i.e., less decay of change).

Aim 2: Investigate theoretical mechanisms through which +Change conditions impact alcohol use (e.g., descriptive drinking norms, drinking to cope with minority stress for LGBTQ students), sexual assault victimization and perpetration (e.g., sexual assault-related norms, sexual assault resistance self-efficacy, hypergender ideology), and bystander intervention (e.g., bystander intervention self-efficacy).

Exploratory Aim: Examine +Change efficacy among LGBTQ subgroups (lesbian, gay, bisexual, trans, non-binary gender, gender queer, queer/questioning, intersex, asexual).

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old
* Current student at university of study
* Valid email address at university of study
* Endorse engaging in heavy episodic drinking at least once in the past month on the screening survey

Exclusion Criteria:

• There are no exclusion criteria other than not meeting inclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3300 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Alcohol use | 3-, 6-, 9-, and 12-months
  Number of drinks will be assessed using the daily drinking questionnaire. Higher scores indicate higher alcohol use.
Changes in Sexual Assault Victimization | 3-, 6-, 9-, and 12-months
  Sexual assault victimization severity will be assessed using a modified version of the Sexual Experiences Survey. Responses are rated on number of times each experience occurred (0, 1, 2, 3+). Higher scores indicate higher sexual assault victimization.
Changes in Bystander Intervention | 3-, 6-, 9-, and 12-months
  Bystander intervention behavior will be assessed using the 44-item Bystander Behavior Scale to assess engaging in bystander behavior with friends. Responses indicate if the participant engaged in each bystander behavior with a friend or not, or if they had no opportunity to engage in the behavior. Higher scores indicate higher bystander intervention behaviors.
Changes in Sexual Assault Perpetration | 3-, 6-, 9-, and 12-months
  Sexual assault perpetration severity will be assessed using a modified version of the Sexual Strategies Survey. Participants check all items that apply. Higher scores indicate higher sexual assault perpetration.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gilmore, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided